CLINICAL TRIAL: NCT00800384
Title: Shockless Implant Evaluation
Acronym: SIMPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-2007
Record Dates: First submitted 2008-11-27; First posted 2008-12-02 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2014-03

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ICD implant without defibrillation testing
  Interventions: Device: Implantable defibrillator
- 2 (Active Comparator): ICD implant with defibrillation testing
  Interventions: Device: Implantable defibrillator

INTERVENTIONS:
Device: Implantable defibrillator — Implantable defibrillator to detect and terminate ventricular arrhythmias
  Other Names: Study is not device specific.; Any market released ICD including cardiac resynchromization therapy (CRT)-Ds can be included.

SUMMARY:
This trial will assess the safety of defibrillator testing and the influence of defibrillation testing on the efficacy of clinical shocks.

The trial will test the hypothesis that implantable cardioverter defibrillator (ICD) implantation without defibrillation testing (DT) is non-inferior to implantation with testing against the composite endpoint of ineffective first appropriate clinical shock or arrhythmic death.

It will also test the hypothesis, that defibrillation testing increases the peri-operative (30 days) complication rate of ICD implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients undergoing initial implant of an ICD or CRT-D device (can be upgrade from a pacemaker)

Exclusion Criteria:

* Patients, who in the opinion of their treating physicians are ineligible for either strategy (DT or no DT)
* Patients on active transplant list
* Patients unwilling to provide informed consent
* Patients not available for follow-up
* Pregnancy or women of child bearing potential not following an effective method of contraception
* Anticipated right sided implantation of the ICD generator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2009-01; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Healey, MD, Principal Investigator — Population Health Research Institute Canada; Stuart Connolly, MD, Study Chair — Population Health Research Institute Canada
Locations (85):
- The Royal Melbourne Hospital, Melbourne, Australia
- Austria (4):
  - Landesklinikum St. Poelten, Sankt Pölten
  - Allgemeines Krankenhaus Wien, Vienna
  - Wilhelminenspital, Vienna
  - Klinikum Wels - Grieskirchen, Wels
- Canada (13):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Jubilee Hospital, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
  - Fleurimont Hospital, Sherbrooke, Quebec
- IKEM - Institut klinicke a experimentalni mediciny, Prague, Czechia
- Tampere University Hospital, Tampere, Finland
- France (5):
  - CHU Grenoble - Hopital Michallon, Grenoble
  - CHRU de Lille, Lille
  - CHRU Nancy Brabois, Nancy
  - CHG de Pau, Pau
  - CHRU Hopital Pontchaillou, Rennes
- Germany (26):
  - Zentralklinik Bad Berka, Bad Berka
  - German Heart Center Berlin, Berlin
  - Heart Center, Bernau
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - University Hospital Bochum Bergmannsheil, Bochum
  - Klinikum Coburg gGmbH, Coburg
  - Klinikum Lippe-Detmold, Detmold
  - Klinikum Dortmund gGmbH, Dortmund
  - University Hospital, Frankfurt
  - University Hospital Heidelberg, Heidelberg
  - Saarland University Hospital, Homburg/Saar
  - Klinikum Kassel, Kassel
  - Krankenhaus Landshut Achdorf, Landshut
  - Medizinische Klinik und Poliklinik I, Leipzig
  - Marienhospital Lünen, Lünen
  - University Hospital of Muenster, Münster
  - Klinikum Nuernberg Sued, Nuremberg
  - Klinikum Oldenburg GmbH, Oldenburg
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - Klinikum der Universitaet Regensburg, Regensburg
  - University of Rostock, Rostock
  - Herzkreislaufzentrum Rotenburg, Rotenburg an der Fulda
  - Krankenhaus der Barmherzigen Brüder, Trier
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - Heinrich Braun Krankenhaus, Zwickau
- Prince of Wales Hospital, Shatin, Hong Kong
- Hungary (3):
  - Hungarian Institute of Cardiology, Budapest
  - Semmelweis University, Cardiovascular Center, Budapest
  - Allami Egeszsegugyi Kozpont (AEK) Hospital, Budapest
- Israel (6):
  - Soroka MC, Beersheba
  - Carmel Medical Center, Haifa
  - Hadassh University Hospital, Mount Scopus, Jerusalem
  - Beilinson Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Netherlands (6):
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Leiden University Medical Center, Leiden
  - Medisch Centrum Haaglanden (MCH) - locatie Westeinde, The Hague
  - Universitair Medisch Centrum, Utrecht
  - Isala Klinieken, Zwolle
- Sorlandet Sykehus HF Kristiansand, Kristiansand, Norway
- Poland (2):
  - Gornoslaskie Centrum Medyczne, Katowice
  - Polsko-Amerykańske Kliniki Serca, Tychy
- Spain (9):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Clinico Y Provincial, Barcelona
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre Madrid, Madrid
  - Hospital La Paz, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital De Navarra, Pamplona
  - H. Clinico Universitario, Valencia
- Karolinska Hospital, Stockholm, Sweden
- Ramathibodi Hospital, Bangkok, Thailand
- United Kingdom (3):
  - St. Peters Hospital, Chertsey
  - Cardiothoracic Centre, Liverpool
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Vamos M, Healey JS, Wang J, Connolly SJ, Mabo P, Van Erven L, Kautzner J, Glikson M, Neuzner J, O'Hara G, Vinolas X, Gadler F, Hohnloser SH. Implantable cardioverter-defibrillator therapy in hypertrophic cardiomyopathy: A SIMPLE substudy. Heart Rhythm. 2018 Mar;15(3):386-392. doi: 10.1016/j.hrthm.2017.11.020. Epub 2017 Nov 20. PMID 29157723
- [Derived] Vamos M, Healey JS, Wang J, Duray GZ, Connolly SJ, van Erven L, Vinolas X, Neuzner J, Glikson M, Hohnloser SH. Troponin levels after ICD implantation with and without defibrillation testing and their predictive value for outcomes: Insights from the SIMPLE trial. Heart Rhythm. 2016 Feb;13(2):504-10. doi: 10.1016/j.hrthm.2015.11.009. Epub 2015 Nov 11. PMID 26569461
- [Derived] Healey JS, Hohnloser SH, Glikson M, Neuzner J, Mabo P, Vinolas X, Kautzner J, O'Hara G, VanErven L, Gadler F, Pogue J, Appl U, Gilkerson J, Pochet T, Stein KM, Merkely B, Chrolavicius S, Meeks B, Foldesi C, Thibault B, Connolly SJ; Shockless IMPLant Evaluation [SIMPLE] investigators. Cardioverter defibrillator implantation without induction of ventricular fibrillation: a single-blind, non-inferiority, randomised controlled trial (SIMPLE). Lancet. 2015 Feb 28;385(9970):785-91. doi: 10.1016/S0140-6736(14)61903-6. Epub 2015 Feb 23. PMID 25715991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was recruited 13 January 2014, last patient was recruited 4 April 2011. All patients were part of the general ICD population at participating sites.
Groups:
- ICD Implant Without Defibrillation Testing: Patients in this arm were implanted with their ICD without having the defibrillation test performed at implant. No VF induction was performed.
- ICD Implant With Defibrillation Testing: Patients in this arm were implanted with their ICD and VF induction was performed followed by shock delivery to test shock efficacy at implant.
Period: Overall Study
Arm/Group | ICD Implant Without Defibrillation Testing | ICD Implant With Defibrillation Testing
Started | 1247 | 1253
Completed | 1206 | 1210
Not Completed | 41 | 43
Not completed — Withdrawal by Subject | 24 | 17
Not completed — Lost to Follow-up | 17 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICD Implant Without Defibrillation Testing | ICD Implant With Defibrillation Testing | Total
Number analyzed (Participants) | 1247 | 1253 | 2500
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.58 (11.51) | 62.98 (11.69) | 62.78 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 244 | 476
  Male | 1015 | 1009 | 2024

OUTCOME MEASURES:

1. Primary Outcome: First Occurrence of the Composite of Failed First Appropriate Clinical Shock From the Implantable Cardioverter Defibrillator (ICD) or Arrhythmic Death
Description: The number of patients having experienced either an appropriate inefficient shock and/or arrhythmic death during the follow-up time frame of 3.1 years is compared between both groups.
Time Frame: Mean follow-up of 3.1 years
Population: All patients were analyzed as per intention to treat. An on treatment analysis was performed in 1190 patients in the group without defibrillation testing and in 1165 patients in the group with defibrillation testing.
Measure: Number; unit: participants
Arm/Group | ICD Implant Without Defibrillation Testing | ICD Implant With Defibrillation Testing
Number analyzed (Participants) | 1247 | 1253
participants | 90 | 104

2. Secondary Outcome: Perioperative Complication Rate
Description: A predefined set of expected complications attributed to defibrillation testing during implant procedure was analyzed in both groups.
Time Frame: 30 days
Population: Perioperative complication rate was assessed in patients undergoing ICD implant. Number of patients having experienced at least one of the predefined complications was assessed.
Measure: Number; unit: participants
Groups:
- ICD Implant With Defibrillation Testing: Patients in this arm were implanted with their ICD and ventricular fibrillation (VF) induction was performed followed by shock delivery to test shock efficacy at implant.
Arm/Group | ICD Implant Without Defibrillation Testing | ICD Implant With Defibrillation Testing
Number analyzed (Participants) | 1236 | 1242
participants | 69 | 81

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first enrollment until last patient last follow-up. Total Follow-up duration 4 years and 10 months. Average follow-up time 3.1 years.
Description: All serious adverse events as per International Standards Organization (ISO) 14155 were collected, regardless whether they were related to the device or protocol. Non serious adverse events were collected without predefining a frequency threshold.
Arm/Group | ICD Implant Without Defibrillation Testing | ICD Implant With Defibrillation Testing
Serious Adverse Events (participants affected / at risk) | 776/1247 | 790/1253
Other Adverse Events (participants affected / at risk) | 625/1247 | 632/1253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD Implant Without Defibrillation Testing (N=1247) | ICD Implant With Defibrillation Testing (N=1253)
PG System (Cardiac disorders) | 2 (2) | 1 (1)
Unable to capture - RV (Cardiac disorders) | 0 (0) | 1 (1)
Unable to convert - Defibrillation (Cardiac disorders) | 2 (2) | 10 (11)
Elevated DFT - Defibrillation (Cardiac disorders) | 0 (0) | 2 (2)
PG system - Therapy (Cardiac disorders) | 1 (1) | 1 (1)
Inappropriate tachy therapy - SVT (Cardiac disorders) | 25 (27) | 25 (30)
Inappropriate tachy therapy - NSR (Cardiac disorders) | 2 (2) | 3 (3)
Inappropriate tachy therapy - Noise (Cardiac disorders) | 0 (0) | 2 (2)
Inappropriate tachy therapy - Other (Cardiac disorders) | 2 (2) | 0 (0)
Early ERI - Random component failure (Cardiac disorders) | 2 (2) | 0 (0)
Early ERI - Consistent with device programming (Cardiac disorders) | 0 (0) | 1 (1)
Early ERI - Premature declaration (Cardiac disorders) | 3 (3) | 4 (4)
Pacemaker-mediated tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
PG System - Patient related (Cardiac disorders) | 0 (0) | 1 (1)
Erosion (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (7)
PG system - Infection (> 30 days post implant) (Infections and infestations) | 24 (29) | 21 (23)
Psychological effect due to device therapy (Psychiatric disorders) | 2 (2) | 1 (1)
Seroma - Pocket (> 30 days post- implant) (Infections and infestations) | 0 (0) | 1 (1)
Migration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Post-surgical wound discomfort (Surgical and medical procedures) | 7 (7) | 2 (2)
Post-surgical pocket hemorrhage (Surgical and medical procedures) | 0 (0) | 4 (4)
Post-surgical infection (<= 30 days post-implant) (Infections and infestations) | 11 (13) | 10 (10)
Adverse reaction - General (Surgical and medical procedures) | 2 (2) | 5 (5)
Adverse reaction - Respiratory (Surgical and medical procedures) | 0 (0) | 6 (6)
Adverse reaction - Hypotension (Surgical and medical procedures) | 1 (1) | 2 (2)
Hemodynamic instability - DFT testing (Surgical and medical procedures) | 0 (0) | 1 (1)
Inadvertent VT/VF (Surgical and medical procedures) | 1 (1) | 5 (5)
Inadvertent SVT (Surgical and medical procedures) | 2 (2) | 3 (3)
Chest pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Hemorrhage (Surgical and medical procedures) | 2 (2) | 5 (5)
Physical trauma (Surgical and medical procedures) | 0 (0) | 2 (2)
Hematoma - Pocket (<=30 days post-implant) (Surgical and medical procedures) | 23 (24) | 31 (31)
Seroma - Pocket (<=30 days post-implant) (Surgical and medical procedures) | 0 (0) | 1 (1)
Thromboembolic events (Surgical and medical procedures) | 6 (7) | 10 (10)
Other - PG system - Procedure (Surgical and medical procedures) | 0 (0) | 2 (2)
Undersensing - RA (Cardiac disorders) | 0 (0) | 1 (1)
Unable to capture - RA (Cardiac disorders) | 2 (2) | 0 (0)
Elevated threshold - RA (Cardiac disorders) | 1 (1) | 2 (2)
Conductor coil fracture - RA (Cardiac disorders) | 1 (1) | 0 (0)
Dislodgment - Unable to capture - RA (Cardiac disorders) | 0 (0) | 3 (4)
Dislodgment - Extracardiac stimulation- RA (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Multiple signs - RA (Cardiac disorders) | 4 (4) | 1 (1)
Dislodgment - No reported signs - RA (Cardiac disorders) | 8 (8) | 8 (9)
Other - Lead (Cardiac disorders) | 2 (2) | 3 (3)
RV - unspecific (Cardiac disorders) | 1 (1) | 1 (1)
Oversensing - RV (Cardiac disorders) | 2 (2) | 0 (0)
Unable to capture - RV (Cardiac disorders) | 7 (7) | 1 (1)
Elevated threshold - RV (Cardiac disorders) | 7 (7) | 6 (6)
Conductor coil fracture - RV (Cardiac disorders) | 0 (0) | 1 (1)
Insulation breach - RV (Cardiac disorders) | 0 (0) | 4 (4)
Electrode damaged - RV (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial perforation post- implant - RV (Cardiac disorders) | 0 (0) | 1 (1)
Impedance < 300 ohms - RV (Cardiac disorders) | 0 (0) | 1 (1)
Impedance > 2000 ohms - RV (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Unable to capture RV (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Elevated threshold -RV (Cardiac disorders) | 7 (7) | 2 (2)
Dislodgment - Oversensing - RV (Cardiac disorders) | 1 (1) | 0 (0)
Dislodgment - Multiple signs - RV (Cardiac disorders) | 3 (3) | 3 (3)
Dislodgment - No reported signs - RV (Cardiac disorders) | 7 (7) | 8 (9)
Unable to capture - LV (Cardiac disorders) | 2 (2) | 3 (3)
Elevated threshold - LV (Cardiac disorders) | 2 (2) | 1 (1)
Extracardiac stimulation - LV (Cardiac disorders) | 4 (4) | 4 (4)
Electrode damaged - LV (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Unable to capture - LV (Cardiac disorders) | 1 (1) | 1 (1)
Dislodgment - Elevated threshold - LV (Cardiac disorders) | 1 (1) | 0 (0)
Dislodgment - Extracardiac stimulation- LV (Cardiac disorders) | 0 (0) | 2 (2)
Dislodgment - Multiple signs - LV (Cardiac disorders) | 1 (1) | 1 (1)
Dislodgment - No reported signs -LV (Cardiac disorders) | 5 (6) | 4 (4)
Oversensing - Defibrillation lead (Cardiac disorders) | 2 (2) | 3 (3)
Undersensing - Defibrillation lead (Cardiac disorders) | 3 (3) | 3 (3)
Elevated DFT - Defibrillation lead (Cardiac disorders) | 1 (1) | 1 (1)
Puncture site hematoma - Procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Pneumothorax - Procedure (Surgical and medical procedures) | 19 (20) | 11 (11)
Renal failure due to contrast media - Procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Pleural effusion - Procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Hemothorax - Procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary venous dissection (Surgical and medical procedures) | 1 (1) | 3 (3)
Myocardial perforation with tamponade (Surgical and medical procedures) | 1 (1) | 2 (2)
AV block (transient) - Procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Pericardial effusion (Surgical and medical procedures) | 7 (8) | 3 (3)
Other - Lead - Procedure (Surgical and medical procedures) | 18 (18) | 18 (18)
Patient CONDITION Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia - unspecific (Cardiac disorders) | 0 (0) | 1 (1)
Bradyarrhythmias - unspecific (Cardiac disorders) | 0 (0) | 1 (1)
1st degree AV block (Cardiac disorders) | 1 (1) | 1 (1)
3rd degree AV block (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Pulseless electrical activity (PEA) (Cardiac disorders) | 2 (2) | 5 (5)
Ventricular tachyarrhythmias - unspecified (Cardiac disorders) | 6 (6) | 7 (8)
Ventricular fibrillation (VF) (Cardiac disorders) | 13 (13) | 7 (8)
Ventricular tachycardia (VT) (Cardiac disorders) | 49 (65) | 38 (57)
Electrical Storm (Cardiac disorders) | 15 (15) | 13 (15)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 5 (5) | 2 (2)
Ventricular flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Tachyarrhythmias - unspecific (Cardiac disorders) | 6 (6) | 2 (2)
Atrial fibrillation (AF) (Cardiac disorders) | 42 (48) | 49 (65)
Atrial flutter (Cardiac disorders) | 13 (17) | 17 (17)
Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 2 (2) | 7 (8)
Atypical Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Premature ventricular contractions (PVC) (Cardiac disorders) | 2 (2) | 4 (4)
Syncope - Heart failure (Cardiac disorders) | 3 (3) | 0 (0)
Dizziness - Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - Heart failure (Cardiac disorders) | 6 (7) | 2 (2)
Dyspnea - Heart failure (Cardiac disorders) | 42 (50) | 41 (50)
Peripheral edema - Heart failure (Cardiac disorders) | 7 (12) | 5 (5)
Pulmonary edema - Heart failure (Respiratory, thoracic and mediastinal disorders) | 23 (26) | 12 (14)
Fatigue - Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Renal insufficiency - Heart failure (Renal and urinary disorders) | 9 (12) | 4 (6)
Dehydration - Heart failure (Cardiac disorders) | 4 (4) | 4 (4)
Gastrointestinal - Heart failure (Gastrointestinal disorders) | 1 (1) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 37 (45) | 42 (62)
Multiple heart failure symptoms (Cardiac disorders) | 145 (212) | 138 (202)
Hypertension - Heart failure (Cardiac disorders) | 2 (2) | 1 (1)
Other- Heart failure patient condition - Cardiovascular (Cardiac disorders) | 7 (7) | 3 (3)
Multi-system failure - Heart failure (Cardiac disorders) | 76 (81) | 57 (63)
Hypotension (Vascular disorders) | 9 (9) | 10 (11)
Hypertension (Vascular disorders) | 3 (3) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 5 (5) | 9 (9)
Cardiac arrest (Cardiac disorders) | 7 (7) | 11 (11)
Myocardial infarction (Cardiac disorders) | 34 (34) | 27 (29)
Coronary Artery Disease (Vascular disorders) | 83 (103) | 46 (63)
Vascular disease - unspecific (Vascular disorders) | 5 (5) | 6 (8)
Peripheral vascular disease (Vascular disorders) | 36 (55) | 37 (62)
Valve related - unspecific (Cardiac disorders) | 13 (13) | 13 (15)
Aortic stenosis (Vascular disorders) | 2 (2) | 4 (4)
Mitral stenosis (Cardiac disorders) | 1 (1) | 1 (2)
Mitral regurgitation (Cardiac disorders) | 3 (3) | 2 (2)
Syncope (General disorders) | 26 (28) | 37 (41)
Dizziness (General disorders) | 8 (8) | 2 (2)
Chest pain - Ischemic (Cardiac disorders) | 20 (25) | 21 (24)
Chest pain - Other (General disorders) | 22 (23) | 19 (22)
Dyspnea (General disorders) | 9 (9) | 9 (9)
Palpitations (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 0 (0)
Other- Patient condition - Cardiovascular (General disorders) | 1 (1) | 1 (1)
Thromboembolic events - unspecific (Vascular disorders) | 0 (0) | 1 (1)
Transient ischemic attack (TIA) (Vascular disorders) | 9 (9) | 12 (12)
Cerebrovascular accident (CVA) (Vascular disorders) | 33 (34) | 23 (26)
Deep vein thrombosis (DVT) (Vascular disorders) | 2 (2) | 1 (1)
Pulmonary embolism (PE) (Vascular disorders) | 6 (6) | 6 (6)
Distal thromboemboli (Vascular disorders) | 8 (8) | 8 (10)
Intracardiac thrombus (Vascular disorders) | 1 (1) | 0 (0)
Procedure related complication other than implant procedure (Surgical and medical procedures) | 16 (21) | 12 (12)
Pericardial effusion - Unrelated to procedure (Surgical and medical procedures) | 2 (2) | 5 (5)
Pericarditis (Surgical and medical procedures) | 0 (0) | 1 (1)
Hematoma (Surgical and medical procedures) | 9 (9) | 5 (5)
Hemorrhage (Surgical and medical procedures) | 6 (7) | 5 (6)
Adverse reaction - Allergic reaction (Immune system disorders) | 3 (3) | 2 (2)
Vasovagal reaction (Vascular disorders) | 3 (3) | 2 (2)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 24 (37) | 15 (25)
WHOLE BODY (General disorders) | 1 (1) | 0 (0)
Death - Reason unspecified (General disorders) | 46 (46) | 50 (50)
Systemic infection (Infections and infestations) | 46 (52) | 36 (40)
Fever (General disorders) | 9 (10) | 3 (3)
Physical trauma (General disorders) | 29 (32) | 37 (42)
Abnormal laboratory values (Blood and lymphatic system disorders) | 8 (8) | 8 (8)
Hematological (Blood and lymphatic system disorders) | 19 (24) | 15 (17)
Neurological (Nervous system disorders) | 15 (17) | 18 (20)
Gastrointestinal (Gastrointestinal disorders) | 95 (132) | 115 (147)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 94 (123) | 95 (115)
Genitourinary (Renal and urinary disorders) | 26 (33) | 38 (46)
Renal (Renal and urinary disorders) | 54 (61) | 41 (52)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 41 (46) | 34 (38)
Psychological (Psychiatric disorders) | 11 (12) | 14 (17)
Integumentary (Skin and subcutaneous tissue disorders) | 20 (23) | 10 (10)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 31 (39) | 23 (25)
Endocrine (Endocrine disorders) | 25 (28) | 32 (35)
Immune (Immune system disorders) | 3 (3) | 3 (3)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 61 (81) | 60 (91)
Multi-system failure (General disorders) | 7 (7) | 12 (12)
(General disorders) | 13 (14) | 14 (15)
Adverse drug reaction (General disorders) | 14 (14) | 13 (13)
(General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICD Implant Without Defibrillation Testing (N=1247) | ICD Implant With Defibrillation Testing (N=1253)
PG System (Cardiac disorders) | 1 (1) | 0 (0)
Oversensing - RA (Cardiac disorders) | 1 (1) | 0 (0)
Other - PG system (Cardiac disorders) | 3 (3) | 0 (0)
Unable to convert - Defibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Elevated DFT - Defibrillation (Cardiac disorders) | 0 (0) | 3 (3)
PG system - Therapy (Cardiac disorders) | 1 (1) | 1 (1)
Inappropriate AV Delay (Cardiac disorders) | 1 (1) | 0 (0)
Inappropriate tachy therapy - SVT (Cardiac disorders) | 20 (23) | 22 (33)
Inappropriate tachy therapy - NSR (Cardiac disorders) | 4 (4) | 6 (6)
Inappropriate tachy therapy - Noise (Cardiac disorders) | 0 (0) | 2 (2)
Inappropriate tachy therapy - Other (Cardiac disorders) | 4 (4) | 1 (1)
Early ERI - Premature declaration (Cardiac disorders) | 1 (1) | 0 (0)
Pacemaker-mediated tachycardia (Cardiac disorders) | 6 (6) | 3 (4)
PG system - Diagnosis (Cardiac disorders) | 1 (1) | 0 (0)
Inability to maintain telemetry (Cardiac disorders) | 0 (0) | 5 (5)
PG System - Patient related (Cardiac disorders) | 6 (6) | 3 (3)
PG system - Infection (> 30 days post implant) (Infections and infestations) | 5 (5) | 3 (3)
Psychological effect due to device therapy (Psychiatric disorders) | 3 (4) | 3 (3)
Hematoma - Pocket (> 30 days post implant) (Surgical and medical procedures) | 2 (2) | 0 (0)
Migration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Post-surgical wound discomfort (Surgical and medical procedures) | 20 (20) | 21 (24)
Post-surgical pocket hemorrhage (Surgical and medical procedures) | 2 (2) | 2 (2)
Post-surgical infection (<= 30 days post-implant) (Infections and infestations) | 8 (8) | 4 (5)
Adverse reaction - General (General disorders) | 6 (6) | 2 (2)
Adverse reaction - Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Adverse reaction - Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Adverse reaction - Hypotension (Surgical and medical procedures) | 3 (3) | 4 (4)
Vasovagal (Surgical and medical procedures) | 5 (5) | 2 (2)
Hemodynamic instability - DFT testing (Surgical and medical procedures) | 0 (0) | 2 (2)
Inadvertent VT/VF (Cardiac disorders) | 1 (1) | 2 (2)
Inadvertent SVT (Cardiac disorders) | 5 (5) | 4 (4)
Chest pain (General disorders) | 1 (1) | 1 (1)
Hemorrhage (Surgical and medical procedures) | 1 (1) | 1 (1)
Physical trauma (Surgical and medical procedures) | 6 (6) | 7 (9)
Hematoma - Pocket (<=30 days post-implant) (Surgical and medical procedures) | 60 (61) | 51 (51)
Seroma - Pocket (<=30 days post-implant) (Surgical and medical procedures) | 4 (4) | 2 (2)
Thromboembolic events (Surgical and medical procedures) | 3 (3) | 10 (10)
Other - PG system - Procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Oversensing - RA (Cardiac disorders) | 3 (3) | 2 (2)
Undersensing - RA (Cardiac disorders) | 1 (1) | 2 (2)
Unable to capture - RA (Cardiac disorders) | 1 (1) | 3 (3)
Elevated threshold - RA (Cardiac disorders) | 6 (6) | 10 (10)
Extracardiac stimulation - RA (Cardiac disorders) | 0 (0) | 1 (1)
Electrode damaged - RA (Cardiac disorders) | 1 (1) | 0 (0)
Impedance > 2000 ohms - RA (Cardiac disorders) | 1 (1) | 1 (1)
Dislodgment - Unable to capture - RA (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Elevated threshold - RA (Cardiac disorders) | 1 (1) | 0 (0)
Dislodgment - Extracardiac stimulation- RA (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Multiple signs - RA (Cardiac disorders) | 1 (1) | 1 (1)
Dislodgment - No reported signs - RA (Cardiac disorders) | 1 (1) | 3 (3)
Other - Lead (Cardiac disorders) | 4 (4) | 8 (9)
Oversensing - RV (Cardiac disorders) | 3 (3) | 1 (1)
Unable to capture - RV (Cardiac disorders) | 0 (0) | 1 (1)
Elevated threshold - RV (Cardiac disorders) | 16 (16) | 15 (15)
Conductor coil fracture - RV (Cardiac disorders) | 0 (0) | 1 (1)
Impedance < 300 ohms - RV (Cardiac disorders) | 1 (1) | 0 (0)
Dislodgment - Elevated threshold -RV (Cardiac disorders) | 0 (0) | 2 (2)
Dislodgment - Multiple signs - RV (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - No reported signs - RV (Cardiac disorders) | 1 (1) | 0 (0)
Unable to capture - LV (Cardiac disorders) | 4 (4) | 1 (1)
Elevated threshold - LV (Cardiac disorders) | 19 (20) | 21 (21)
Extracardiac stimulation - LV (Cardiac disorders) | 32 (41) | 36 (45)
Electrode damaged - LV (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Unable to capture - LV (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Elevated threshold - LV (Cardiac disorders) | 0 (0) | 1 (1)
Dislodgment - Multiple signs - LV (Cardiac disorders) | 1 (1) | 1 (1)
Dislodgment - No reported signs -LV (Cardiac disorders) | 3 (3) | 1 (1)
Defibrillation lead (Cardiac disorders) | 1 (1) | 1 (1)
Oversensing - Defibrillation lead (Cardiac disorders) | 2 (2) | 2 (2)
Undersensing - Defibrillation lead (Cardiac disorders) | 0 (0) | 1 (1)
Elevated DFT - Defibrillation lead (Cardiac disorders) | 2 (2) | 2 (2)
Arterial perforation - Procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Pneumothorax - Procedure (Surgical and medical procedures) | 2 (2) | 4 (4)
Renal failure due to contrast media - Procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Pleural effusion - Procedure (Surgical and medical procedures) | 4 (4) | 4 (4)
Coronary venous dissection (Surgical and medical procedures) | 8 (8) | 3 (3)
AV block (transient) - Procedure (Surgical and medical procedures) | 3 (3) | 0 (0)
Pericardial effusion (Surgical and medical procedures) | 1 (1) | 2 (2)
Other - Lead - Procedure (Surgical and medical procedures) | 23 (24) | 27 (27)
Patient CONDITION Cardiovascular (Cardiac disorders) | 1 (1) | 1 (1)
Bradyarrhythmias - unspecific (Cardiac disorders) | 2 (2) | 0 (0)
1st degree AV block (Cardiac disorders) | 2 (2) | 0 (0)
2nd degree AV block (Cardiac disorders) | 2 (2) | 0 (0)
3rd degree AV block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 4 (4)
Chronotropic incompetence (Cardiac disorders) | 3 (3) | 2 (2)
Ventricular tachyarrhythmias - unspecified (Cardiac disorders) | 3 (3) | 2 (2)
Ventricular fibrillation (VF) (Cardiac disorders) | 2 (7) | 5 (5)
Ventricular tachycardia (VT) (Cardiac disorders) | 23 (25) | 33 (39)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 7 (10) | 14 (17)
Accelerated idiopathic rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Tachyarrhythmias - unspecific (Cardiac disorders) | 6 (6) | 1 (1)
Atrial fibrillation (AF) (Cardiac disorders) | 45 (49) | 43 (49)
Atrial flutter (Cardiac disorders) | 12 (13) | 6 (6)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 4 (4) | 5 (6)
Premature ventricular contractions (PVC) (Cardiac disorders) | 7 (7) | 5 (6)
Syncope - Heart failure (Cardiac disorders) | 3 (3) | 0 (0)
Dizziness - Heart failure (Cardiac disorders) | 4 (5) | 2 (4)
Chest pain - Heart failure (Cardiac disorders) | 1 (1) | 4 (4)
Dyspnea - Heart failure (Cardiac disorders) | 34 (37) | 29 (29)
Peripheral edema - Heart failure (Cardiac disorders) | 15 (15) | 11 (11)
Pulmonary edema - Heart failure (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Fatigue - Heart failure (Cardiac disorders) | 6 (6) | 6 (8)
Renal insufficiency - Heart failure (Renal and urinary disorders) | 3 (3) | 2 (2)
Dehydration - Heart failure (Cardiac disorders) | 2 (2) | 1 (1)
Weight gain - Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 10 (10) | 5 (5)
Multiple heart failure symptoms (Cardiac disorders) | 31 (34) | 33 (39)
Hypertension - Heart failure (Cardiac disorders) | 2 (2) | 0 (0)
Other- Heart failure patient condition - Cardiovascular (Cardiac disorders) | 5 (5) | 2 (2)
Hypotension (Vascular disorders) | 22 (22) | 19 (19)
Hypertension (Vascular disorders) | 9 (9) | 15 (18)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 18 (19) | 14 (14)
Vascular disease - unspecific (Vascular disorders) | 6 (6) | 4 (4)
Peripheral vascular disease (Vascular disorders) | 12 (12) | 5 (7)
Valve related - unspecific (Cardiac disorders) | 2 (2) | 1 (1)
Syncope (General disorders) | 43 (48) | 27 (31)
Dizziness (General disorders) | 26 (30) | 36 (38)
Chest pain - Ischemic (Cardiac disorders) | 10 (11) | 11 (11)
Chest pain - Other (General disorders) | 17 (28) | 19 (23)
Dyspnea (General disorders) | 19 (20) | 12 (12)
Palpitations (General disorders) | 12 (13) | 9 (9)
Fatigue (General disorders) | 10 (10) | 6 (6)
Multiple Symptoms (General disorders) | 1 (1) | 4 (4)
Thromboembolic events - unspecific (Vascular disorders) | 2 (2) | 1 (1)
Transient ischemic attack (TIA) (Vascular disorders) | 5 (5) | 3 (3)
Cerebrovascular accident (CVA) (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (DVT) (Vascular disorders) | 0 (0) | 1 (1)
Distal thromboemboli (Vascular disorders) | 4 (4) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 3 (3) | 2 (2)
Procedure related complication other than implant procedure (Surgical and medical procedures) | 7 (10) | 4 (4)
Pericardial effusion - Unrelated to procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Pericarditis (Surgical and medical procedures) | 1 (2) | 0 (0)
Hematoma (Surgical and medical procedures) | 5 (5) | 3 (3)
Hemorrhage (Surgical and medical procedures) | 2 (2) | 0 (0)
Adverse reaction - Allergic reaction (Immune system disorders) | 6 (6) | 7 (7)
Vasovagal reaction (Vascular disorders) | 5 (5) | 5 (5)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
WHOLE BODY (General disorders) | 0 (0) | 2 (2)
Systemic infection (Infections and infestations) | 17 (18) | 3 (3)
Fever (General disorders) | 8 (8) | 1 (1)
Physical trauma (General disorders) | 41 (46) | 30 (31)
Abnormal laboratory values (Blood and lymphatic system disorders) | 14 (15) | 5 (5)
Hematological (Blood and lymphatic system disorders) | 18 (20) | 12 (14)
Neurological (Nervous system disorders) | 16 (17) | 16 (24)
Gastrointestinal (Gastrointestinal disorders) | 49 (62) | 56 (64)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 48 (54) | 59 (68)
Genitourinary (Renal and urinary disorders) | 38 (49) | 28 (32)
Renal (Renal and urinary disorders) | 20 (22) | 14 (14)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 51 (61) | 49 (52)
Psychological (Psychiatric disorders) | 8 (8) | 14 (14)
Integumentary (Skin and subcutaneous tissue disorders) | 30 (32) | 30 (32)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 53 (61) | 49 (53)
Endocrine (Endocrine disorders) | 41 (49) | 38 (44)
Immune (Immune system disorders) | 2 (2) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (17) | 13 (15)
(General disorders) | 16 (17) | 21 (23)
Adverse drug reaction (General disorders) | 26 (30) | 25 (27)
(General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less